CLINICAL TRIAL: NCT06388031
Title: A Multicenter, Single-Arm Pilot Study of Immune Checkpoint Inhibitors in Patients With Locally Advanced or Metastatic Non-Small-Cell Lung Cancer Who Had Long-Term (Two Years or Longer) Response to First-Line Immunotherapy
Brief Title: ICI Rechallenge for Advanced NSCLC With Long-Term Response to First-Line ICI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Minjiang Chen, Assoc. Prof., Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPTRAL2024v1
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy (Experimental): Immune checkpoint inhibitor (anti-PD/1 or anti-PD-L1) monotherapy
  Interventions: Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Drug: Immune checkpoint inhibitor — Physician's choice immunotherapy with one of the following every 21 days until disease progression or intolerable toxicity or up to 17 cycles:
  * Pembrolizumab 200mg;
  * Tislelizumab 200mg;
  * Camrelizumab 200mg;
  * Toripalimab 240mg.
  Other Names: Keytruda

SUMMARY:
An exploratory phase II trial of immune checkpoint inhibitors (ICIs, anti-PD-1/anti-PD-L1) as second-line treatment with advanced non-small cell lung cancer (NSCLC) who had long-term response to first-line immunotherapy (with or without chemotherapy).

This study aims to evaluate efficacy and safety of ICI rechallenge in long-term responders to prior ICI. Furthermore, it seeks to identify biomarkers capable of predicting the efficacy of immunotherapy and prognosis.

DETAILED DESCRIPTION:
This is a multi-center study. The study plans to include a total of 27 advanced NSCLCs who had benefited from first-line immunotherapy over two years before disease progression.

Participants will receive up to 17 cycles of ICI (anti-PD-1 or anti-PD-L1) monotherapy.

Optional ICI monotherapy regimens include: Pembrolizumab 200mg every 3 weeks, or Tislelizumab 200mg every 3 weeks, or Camrelizumab 200mg every 3 weeks, or Toripalimab 240mg every 3 weeks.

The outcomes including efficacy and safety will be examined. Additionally, peripheral blood samples will be collected before treatment, and at the 6th, 12th, and 24th weeks after treatment initiation to explore biomarkers for immunotherapy. Also it is highly recommended to collect pretreatment tumor tissue from patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a thorough understanding of this study and voluntarily sign an informed consent form (ICF);
2. Age between 18 and 80 years, any gender;
3. Histologically or cytologically confirmed stage III-IV non-small cell lung cancer (NSCLC);
4. Previous treated with first-line immunotherapy (immunotherapeutic agents include currently marketed anti-PD-L1 or anti-PD-1 monoclonal antibodies: pembrolizumab, nivolumab, atezolizumab, durvalumab, tislelizumab, toripalimab, sintilimab, camrelizumab, etc.; investigational drugs not yet marketed need discussion with the study team prior to enrollment; with or without platinum-based doublet chemotherapy) for at least 35 cycles or disease stability confirmed by imaging assessment for at least 2 years, and disease progression;
5. Measurable disease (at least 1 lesion) according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1);
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
7. Adequate organ function:

   Hematology: Absolute neutrophil count (ANC) ≥1500/μL; Platelets ≥100000/μL; Hemoglobin ≥9.0g/dL; Renal: Serum creatinine ≤1.5×ULN or calculated creatinine clearance (CrCl) ≥60 mL/min (using Cock-Gault formula); Hepatic: Total bilirubin ≤1.5 ×ULN or, for subjects with total bilirubin levels >1.5×ULN, direct bilirubin within normal limits; AST (SGOT) and ALT (SGPT) ≤2.5×ULN; Coagulation: International normalized ratio (INR) or prothrombin time (PT), activated partial thromboplastin time (APTT) ≤1.5×ULN;
8. Subjects must be willing and able to comply with study visits, treatment plans, laboratory tests, and other study procedures;
9. Female subjects of childbearing potential and male subjects with female partners of childbearing potential must agree to use highly effective contraception during the study and for 180 days after the last dose of the study drug.

Exclusion Criteria:

1. Received two or more prior systemic therapies;
2. Known sensitive EGFR mutation (EGFR exon19 del or EGFR exon21 L858R) or ALK rearrangement;
3. Symptomatic or progressing CNS metastases, leptomeningeal metastases;
4. History of autoimmune disease, active autoimmune disease, immunodeficiency, or requiring systemic corticosteroid/immunosuppressive therapy; (except: a history of hypothyroidism; well-controlled stable type I diabetes mellitus);
5. Idiopathic pulmonary fibrosis (including interstitial pneumonia), drug-induced pneumonitis, history of (non-infectious) pneumonia/interstitial lung disease requiring steroid therapy;
6. Known active tuberculosis, human immunodeficiency virus (HIV) infection; active hepatitis B (defined as positive HBsAg or positive hepatitis B virus DNA test result above the detection limit) or hepatitis C (defined as known positive HCV antibody result, known quantitative HCV-RNA analysis result above the detection limit) history; other known active infections requiring systemic therapy;
7. Received systemic immunostimulatory therapy within 4 weeks before initiation of study treatment or within 5 half-lives of the drug (whichever is longer);
8. Pregnancy, lactation, planning to become pregnant, or fathering a child during the anticipated duration of the study (from screening visit to 180 days after the last dose of investigational drug);
9. Prior allogeneic tissue/organ transplantation and other conditions unsuitable for immunotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2027-01-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 5 months
  Time from the date of treatment start to date of disease progression met by RECIST 1.1 or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | 24 months
  Time from the date of treatment start to date of death from any cause.
Objective Response Rate (ORR) | 5 months
  Proportion of patients with complete and partial responses to immunotherapy according to RECIST 1.1.
Progression Free Survival 2 (PFS 2) | 12 months
  Time from the date of treatment start to the date of disease progression or death after initiation of subsequent anti-tumor therapy.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 24 months
  Evaluate adverse events of any cause, treatment-related adverse events, immune-mediated adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Minjiang Chen, MD., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The result of the study and all the supporting informations will be shared in the form of publishing article.